CLINICAL TRIAL: NCT05553782
Title: Therapeutic Drug Screening Using a Novel Implantable Microdevice (IMD) in Head and Neck Cancers: a Window of Opportunity Study
Brief Title: Drug Screening Using Novel IMD in Salivary and Head and Neck Cancers
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Adenoid Cystic Carcinoma Research Foundation (Other)
Responsible Party: Principal Investigator, Glenn J. Hanna, M.D., Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-381
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Salivary Gland Cancer; Adenoid Cystic Carcinoma of the Salivary Gland; Squamous Cell Carcinoma of Head and Neck; Head and Neck Cancer
Keywords: Salivary Gland Cancer; Adenoid Cystic Carcinoma of the Salivary Gland; Implantable Microdevice IMD; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- IMD PLACEMENT + SURGICAL RESECTION + ADJUVANT TREATMENT ARM (Experimental): Newly diagnosed, localized head and neck cancers undergoing surgical resection
  * Interventional radiology guided IMD placement
  * Planned oncologic resection with IMD retrieval 3-5 days after placement
  * Standard of care adjuvant treatment
  * Tumor specimen analysis for local drug response and molecular analysis
  Interventions: Combination Product: Implantable Microdevice (IMD)

INTERVENTIONS:
Combination Product: Implantable Microdevice (IMD) — * Percutaneous CT image-guided placement of the microdevice(s). At least one, and up to 3, devices will be placed in each tumor.
  * Drugs will be released from the microdevice into local tumor tissues. The duration of drug release will be for a period of 3-5 days while the microdevice is in the tumor prior to retrieval. The local tissue is retrieved along with the microdevice and no residual drug will remain.
  * Each microdevice harbors up to 20 drugs and/or drug combinations relevant to the treatment of head and neck cancer. The drugs used will include some standard agents approved by the Food and Drug Administration (FDA) for treatment of different types of cancers, or drugs classes under investigational.
  * Drugs may include all or a subset of the following which each may be tested as single agents or in any number of combinations including, but not limited to: Lenvatinib, Axitinib, All trans retinoic acid (ATRA), Venetoclax, Pembrolizumab, Cisplatin, Carboplatin, Vinorelbine

SUMMARY:
This research study is studying the effect of different drugs as possible treatments for salivary and other head and neck cancers/

The name of the study intervention involved in this study is:

-- implantable microdevice

DETAILED DESCRIPTION:
This window-of-opportunity pilot study will assess the safety and feasibility of using an implantable microdevice (IMD) to efficiently measure local intratumor response to multiple drugs within previously untreated head and neck cancer patients undergoing definitive oncologic resection.

* This research study is a Pilot Study, which is the first-time investigators are examining this study device in salivary and head and neck cancers. The placement and removal of the microdevice is being tested for the first time in this type of cancer.
* This research study involves drugs that are released by a small implantable microdevice (IMD) as small as the tip of a needle, that is inserted into the tumor and is then removed 3-5 days later during surgery.
* The microdevice can hold up to 20 drugs alone or in combinations in very small concentrations that are able to access the cancer through small pores in the device. When the device is removed along with the cancer at the time of surgery, it will be evaluated to understand which drug(s) may be effective to treat these cancers.

It is expected that about 30 people will take part in this research study.

The U.S. Food and Drug Administration (FDA) has not approved the microdevice a treatment for any disease.

AACRF, a research foundation, is supporting this research study by providing funding for the research study, the study drugs and study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed head and neck cancer (salivary or ACC type, or squamous cell carcinoma) without evidence of recurrent, metastatic or advanced, incurable disease undergoing definitive surgical management; any stage disease is permitted (American Joint Committee on Cancer 2017 8th edition).
* Age 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* A measurable primary tumor site both clinically and radiologically measuring at least 1 x 1 cm.

  - Patients must be deemed medically fit to undergo both percutaneous and surgical procedures by their treating head and neck surgeon and medical oncologist.
* Participants will undergo laboratory testing within 7 days prior to the microdevice placement: they are required to have a platelet count ≥50,000/mcL, PT/INR <2, and aPTT <1.5x upper limit of normal.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 14 days
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit the safety of a biopsy and/or surgery.
* Pregnant women are excluded from this study because of the possible increased dose of radiation from imaging associated with the device placement and the potential risk to the pregnancy of the surgery/device placement.
* Uncorrectable bleeding or coagulation disorder known to cause increased risk with surgical or percutaneous biopsy procedures. If the patient is on systemic anticoagulation, this should be discussed with the overall PI and treating surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or Higher Treatment-Related Toxicity Rate | AE assessed on post-operative visit, which take placed between 7-14 days after the surgical procedure.
  All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.

SECONDARY OUTCOMES:
Pharmacodynamic (PD) | Screening Period 1 day
  Pharmacodynamics reported based on dose/exposure efficacy and safety relationships, there are no clinically significant differences in efficacy and safety between pembrolizumab doses of 200 mg or 2 mg/kg every 3 weeks in patients with melanoma or NSCLC.
Evaluate the likelihood of independent drug or combination response/failure in this pilot population to determine the appropriateness of nominating therapies for further clinical investigation | through study completion, an average of 1 year
Tumor Response | through study completion, an average of 1 year
  Tumor molecular profiling using a commercially available assay (CARIS® MI Profile) will be performed on pathology material from resection sent for permanent processing using cut unstained tissue slides, in post-operative visit up 14 days
Gene Expression Level | through study completion, an average of 1 year
  Tumor molecular profiling using a commercially available assay (CARIS® MI Profile) will be performed on pathology material from resection sent for permanent processing using cut unstained tissue slides, in post-operative visit up to 14 Days
Changes in Tumor Metabolism | through study completion, an average of 1 year
  Tumor molecular profiling using a commercially available assay (CARIS® MI Profile) will be performed on pathology material from resection sent for permanent processing using cut unstained tissue slides, in post-operative visit up to 14 Days
Biomarker levels | through study completion, an average of 1 year
  For hypothesis-generating biomarker discovery, genome-wide approaches looking at both established and novel candidate biomarkers may be able to identify new biomarkers in head and neck cancer

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Hanna, M.D, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu